CLINICAL TRIAL: NCT02470949
Title: Influence of a Monopoly Game on Subtle Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Alabama at Birmingham (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 14-0719
Record Dates: First submitted 2014-10-28; First posted 2015-06-12 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Eating Behavior
Keywords: body weight; Hispanics; Energy Intake; Social Status
MeSH Terms: conditions — Obesity; Feeding Behavior; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Social Status (Experimental): Low Social Status Condition in Monopoly Game.
  Interventions: Behavioral: Low Social Status
- High Social Status (Experimental): High Social Status Condition in Monopoly Game
  Interventions: Behavioral: High Social Status

INTERVENTIONS:
Behavioral: Low Social Status — The participants will be randomized to the Low Social Status Condition. On their second visit, they will undergo the condition in which they were not randomized to on their first visit.
  Arms: Low Social Status
Behavioral: High Social Status — The participants will be randomized to the High Social Status Condition. On their second visit, they will undergo the condition in which they were not randomized to on their first visit.
  Arms: High Social Status

SUMMARY:
This project will investigate the influence of experimentally manipulated perceived social standing on eating behavior and obesity risk.

DETAILED DESCRIPTION:
The scope of work outlined in this proposal will investigate experimentally manipulated social status on acute eating behavior, energy intake, and risk for obesity. This will be accomplished using a randomized, crossover design to place young adults in experimental high and low social status conditions. At visit 1, participants will complete baseline measurements, and then consume a standardized breakfast. In order to control for the influence of stress on eating behavior in both conditions, the participants will participate in the Stroop Test, a test known to induce stress in individuals, following breakfast. Using a computerized randomization scheme, each participant will be randomized to either the low or high social status condition (½ will receive high first; ½ will receive low first) and will receive the packet of rules and instructions for their respective condition. The participants will play Monopoly for up to 2 hours with another player they have not previously met. At the end of the game, the high social status player will be told that they won, and the low social status player will be told that they lost. The participants will participate in the Stroop Test again. Then the investigators will take the players into the Children's Eating Laboratory, where a buffet ad libitum lunch will be served in separate rooms. The participants will have 30 minutes to consume their lunch and plate waste will be measured to assess each participant's dietary intake. There will be a 4-week washout period and the second visit will be exactly like the first, except that they will participate in the alternate social status condition. The investigators will evaluate whether there was within-subject variation in dietary intakes based upon which social status condition they were placed in.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19-25
* Self-identified Hispanic ethnicity
* Born in the United States
* Body Mass Index (BMI) ≥18.5 and ≤30 kg/m2
* A score on the MacArthur scale of subjective social status ≥3 and ≤8
* No self-report of acute or chronic disease (heart disease, diabetes, gastrointestinal disorders in particular)
* No plans for extended travel (>1 week) within the next 2 months
* No current tobacco use
* Capable and willing to give informed consent, understand inclusion criteria, and accept the randomized assignment

Exclusion Criteria:

* Never played monopoly before
* Not born in the United States
* Strict dietary restrictions (vegan, vegetarian, gluten-free, dairy-free/lactose intolerant, nut-allergies)
* Participation in any weight reduction program, weight-loss diet, or other special diet within the previous 3 months
* Weight loss or gain of ≥10 pounds in the past 6 months for any reason except post-partum weight loss
* Currently taking medication that suppresses or stimulates appetite
* Current smoker or quit smoking less than 6 months prior
* Any major disease, including:

  * Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
  * Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
  * Diagnosis of cardiovascular disease
  * Gastrointestinal disease, including inflammatory bowel disease that has required treatment in the past year, celiac disease, recent of significant abdominal surgery
  * Active renal disease
  * Lung disease such as chronic obstructive airway disease requiring use of oxygen
  * Diagnosis of diabetes (type 1 or type 2)
* Uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in the opinion of the investigators, would impede conduct of the trial or completion of procedures
* A score on the Brief Symptom Inventory (BSI) (Derogatis & Melisaratos, 1983) that exceeds the 90th percentile
* History of or current eating disorders, or an Eating Attitudes Test (EAT-26) score >20.
* Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; another household member is a participant or staff member in the trial; unwilling to accept social status assignment by randomization; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating university before visits are completed; unable to walk 0.25 mile in 10 minutes.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months.
* A recent or ongoing problem with drug abuse or addiction.
* Excessive alcohol intake, either acute or chronic, defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months; or 3) other evidence available to clinic staff.
* Not willing to be randomized to any of the two experimental conditions.
* Pregnancy and childbearing: currently pregnant or less than 3 months post-partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the course of the trial; unwilling to take adequate contraceptive measures if potentially fertile.
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cardel, PhD, RD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver-Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the greater Denver, Colorado area in 2015 via flyers, online ads, television, and participant referrals.
Groups:
- Low Social Status, Then High Social Status: Low Social Status Condition in Monopoly Game during the first intervention period and High Social Status Condition in Monopoly Game during the second intervention period (after washout period).
- High Social Status, Then Low Social Status: High Social Status Condition in Monopoly Game during the first intervention period and Low Social Status Condition in Monopoly Game during the second intervention period (after washout period).
Period: First Intervention
Arm/Group | Low Social Status, Then High Social Status | High Social Status, Then Low Social Status
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Washout Period for a Minimum of 4 Weeks
Arm/Group | Low Social Status, Then High Social Status | High Social Status, Then Low Social Status
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Low Social Status, Then High Social Status | High Social Status, Then Low Social Status
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: High Social Status Condition in Monopoly Game and Low Social Status Condition in Monopoly Game
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.8 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Calories Consumed Following the Experimental Manipulation
Description: The participants will be provided with an ad libitum lunch for 20 minutes following the completion of their manipulated social status condition.
Time Frame: Administered 30 days apart
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- Low Social Status: Low Social Status Condition in Monopoly Game.
  Manipulated Social Status: The participants will be randomized to either the Low Social Status Condition or the High Social Status condition. On their second visit, they will undergo the condition in which they were not randomized to on their first visit.
- High Social Status: High Social Status Condition in Monopoly Game
  Manipulated Social Status: The participants will be randomized to either the Low Social Status Condition or the High Social Status condition. On their second visit, they will undergo the condition in which they were not randomized to on their first visit.
Arm/Group | Low Social Status | High Social Status
Number analyzed (Participants) | 8 | 7
kcal | 647.5 (252.8) | 520.9 (231.2)

2. Primary Outcome: The Macronutrient Composition of Foods Consumed
Description: The participants will be provided with an ad libitum lunch for 30 minutes following the completion of their manipulated social status condition.
Time Frame: Administered 30 days apart
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Low Social Status | High Social Status
Number analyzed (Participants) | 8 | 7
grams
  Total Fat | 22.4 (8.6) | 17.0 (9.1)
  Total Carbohydrate | 89.3 (37.1) | 75.4 (29.9)
  Total Sugar | 35.4 (19.2) | 30.9 (14.0)
  Added Sugar | 24.2 (14.8) | 19.3 (9.7)
  Fiber | 6.2 (3.0) | 5.9 (2.4)

3. Primary Outcome: Percent of Calories Consumed Following the Experimental Manipulation
Description: as for outcome 2
Time Frame: Administered 30 days apart
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Low Social Status | High Social Status
Number analyzed (Participants) | 8 | 7
percent
  Percent of Calories from Fat | 30.5 (3.3) | 27.9 (3.5)
  Percent of Calories from Carbohydrate | 54.6 (5.4) | 58.0 (6.0)
  Percent of Calories from Saturated Fat | 14.3 (1.7) | 12.3 (1.9)
  Percent of Energy Needs | 0.39 (0.13) | 0.31 (0.10)

ADVERSE EVENTS:
Description: Not all participants completed both interventions.
Arm/Group | Low Social Status | High Social Status
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No